CLINICAL TRIAL: NCT07225127
Title: Comparison of Intravesical Therapy and Surgery as Treatment Options for Bladder Cancer 2
Acronym: CISTO2
Status: Recruiting | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, John Gore, Vice Chair of Research, Professor, School of Medicine: Urology, University of Washington
Other Study IDs: RG1126118; R01CA289268 (NIH)
Record Dates: First submitted 2025-11-03; First posted 2025-11-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-10

CONDITIONS: Bladder Cancer; Recurrent Bladder Cancer; Non-muscle Invasive Bladder Cancer (NMIBC)
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients who have selected radical cystectomy: Patients with a diagnosis of recurrent high-grade NMIBC who have selected radical cystectomy
- Patients who have selected bladder-sparing therapy: Patients with a diagnosis of recurrent high-grade NMIBC who have selected bladder-sparing therapy (BST)
- Caregivers of patients who have selected radical cystectomy: Caregivers of patients with a diagnosis of recurrent high-grade NMIBC who have selected radical cystectomy
- Caregivers of patients who have selected bladder-sparing therapy: Caregivers of patients with a diagnosis of recurrent high-grade NMIBC who have selected bladder-sparing therapy (BST)

SUMMARY:
Bladder cancer is the most common urinary tract cancer and the 6th most common cancer in the US. Yet bladder cancer research is underfunded relative to other common cancers. As a result, bladder cancer care is prone to evidence gaps that produce decision uncertainty for both patients and clinicians. The Comparison of Intravesical Therapy and Surgery as Treatment Options for Bladder Cancer Study 2 (CISTO2) has the potential to fill these critical evidence gaps, change care pathways for the management of NMIBC (non-muscle-invasive bladder cancer), and provide for personalized, patient-centered care. The purpose of CISTO2 is to conduct a large prospective study that directly compares the impact of bladder sparing therapies versus bladder removal in recurrent high-grade NMIBC patients on financial toxicity, clinical outcomes and patient and caregiver experience using standardized patient-reported outcomes (PROs).

ELIGIBILITY:
Inclusion Criteria:

1. Adult 18 years of age or older; and
2. Presenting with high-grade NMIBC established by anatomic pathology as tumor stage classification Tis, Ta, or T1, and with:

   1. Pathology documentation from any hospital/clinic/medical center
   2. More than 50% urothelial carcinoma component in the specimen; and
3. History of high-grade NMIBC established by anatomic pathology as tumor stage classification Tis, Ta, or T1; and
4. In the previous 12 months, received at least one instillation of any intravesical agent (induction or maintenance) or one administration of systemic therapy for NMIBC treatment.

Exclusion Criteria:

1. Any plasmacytoid or small cell (neuroendocrine) component in the pathology (past or current presentation);
2. Previous history of cystectomy or radiation therapy for bladder cancer;
3. Previous history of muscle-invasive bladder cancer or metastatic bladder cancer;
4. Untreated or current urinary tract urothelial carcinoma outside of the bladder (e.g. ureters, renal pelvis, penile urethra for males, urethra for females). Urinary tract cancer outside of the bladder treated more than 2 years ago is not an exclusion;
5. Incarcerated in a detention facility or in police custody at baseline/screening (patients wearing a monitoring device can be enrolled);
6. Contraindication to radical cystectomy (e.g., ASA of 4, patient not considered a radical cystectomy candidate due to comorbidity);
7. Contraindication to BST (i.e., intolerant of all intravesical and intravenous medical therapies);
8. Unable to provide written informed consent in English;
9. Unable to be contacted for research surveys;
10. Planning to participate in a blinded interventional clinical trial for NMIBC such that details about treatment or therapy received will be unavailable for data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of recurrent high-grade NMIBC who are considering their next treatment will be approached for participation in this observational study in addition to their caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 408 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Patient-reported financial toxicity as measured by the COmprehensive Score for financial Toxicity (COST) | 12 months after enrollment
  The primary outcome of patient-reported financial toxicity is measured by the COST measure. The questionnaire consists of 11 items, each scored on a 5-point Likert scale from zero to four. After reversing some items as indicated in the scoring manual (by reversing the sign on the original zero to four score and adding four), all item response scores are summed into a single financial toxicity score ranging from 0 to 44, with higher scores indicating less financial toxicity. Item nonresponse is accounted for by summing the items answered, multiplying by the total number of items in the scale, and then dividing by the number of items that were actually answered.

SECONDARY OUTCOMES:
Patient-reported financial toxicity as measured by the COmprehensive Score for financial Toxicity (COST) | 24 months after enrollment
  Patient-reported financial toxicity is measured by the COST measure. The questionnaire consists of 11 items, each scored on a 5-point Likert scale from zero to four. After reversing some items as indicated in the scoring manual (by reversing the sign on the original zero to four score and adding four), all item response scores are summed into a single financial toxicity score ranging from 0 to 44, with higher scores indicating less financial toxicity. Item nonresponse is accounted for by summing the items answered, multiplying by the total number of items in the scale, and then dividing by the number of items that were actually answered.
Caregiver self-reported financial distress as measured by the modified Comprehensive Score for Financial Toxicity (COST) | 12 months after enrollment
  Caregiver-reported financial toxicity is measured by the COST measure. The questionnaire consists of 12 items, each scored on a 5-point Likert scale from zero to four. After reversing some items as indicated in the scoring manual (by reversing the sign on the original zero to four score and adding four), all item response scores are summed into a single financial toxicity score ranging from 0 to 44, with higher scores indicating less financial toxicity. Item nonresponse is accounted for by summing the items answered, multiplying by the total number of items in the scale, and then dividing by the number of items that were actually answered.
Patient self-reported financial well-being as measured by the Consumer Financial Protection Bureau (CFPB) Financial Well-Being Scale | 12 months after enrollment
  Patient-reported financial well-being is measured by the CFPB financial well-being scale. The scale consists of 10 items plus 2 questions to assist with scoring. Total response values are converted into an overall financial well-being score between 0 to 100, with higher scores indicating better financial wellness. The financial well-being scores vary based on age and how the questionnaire was administered.
Caregiver self-reported financial well-being as measured by the Consumer Financial Protection Bureau (CFPB) Financial Well-Being Scale | 12 months after enrollment
  Caregiver-reported financial well-being is measured by the CFPB financial well-being scale. The scale consists of 10 items plus 2 questions to assist with scoring. Total response values are converted into an overall financial well-being score between 0 to 100, with higher scores indicating better financial wellness. The financial well-being scores vary based on age and how the questionnaire was administered.
Caregiver self-reported quality of life as measured by the CareGiver Oncology Quality of Life questionnaire (CarGOQol) | 12 months after enrollment
  Caregiver-reported quality of life is measured by the CarGOQol questionnaire. The CarGOQol consists of 29 items, with 5-point Likert response scales, covering 10 domains. The scores for each domain are obtained by calculating the average item score for that domain. The overall score is calculated as the average of the domain scores. A domain score is calculated when more than half of the questions are answered. All domain scores and the overall score are linearly transformed and moralized using a scale of 0 to 100. Higher scores indicate better quality of life for the caregiver.
Patient-reported quality of life as measured by the Physical Function scale of the European Organization for Research and Treatment of Cancer Quality-of-Life-Questionnaire-Core-30 (EORTC QLQ-C30) | 12 months after enrollment
  Patient-reported quality of life is measured by the EORTC QLQ-C30 Physical Function scale. The scale ranges in score from 0 to 100, with higher function scores indicating better health. Scale score is calculated by transforming individual item scores into a 0 to 1 scale, taking the mean, and multiplying by 100. Each scale requires responses for at least 50% of the items to be calculated.
Patient self-reported urinary health as measured by the Bladder Cancer Index urinary summary score | 12 months after enrollment
  Patient-reported urinary health is measured by the Bladder Cancer Index (BCI). The BCI consists of 36 items, with 4- or 5-point Likert response scales, covering 3 primary domains: urinary, bowel, and sexual. For each domain a summary score is constructed from the items used to calculate the two subscale scores (function and bother). Scores are calculated by transforming item responses into a 0 to 100 scale and calculating the mean of the standardized items. Higher scores indicate better health status. To calculate a score, a minimum of 80% completed items is required.
Patient-reported anxiety as measured by the Patient Reported Outcome Measurement Information System (PROMIS) Short Form v1.0 - Anxiety 4a | 12 months after enrollment
  Patient-reported anxiety is measured by the PROMIS Short Form v1.0 - Anxiety 4a. Scores range from 0 to 100, with higher scores indicating greater symptoms. Scores are normalized to a mean of 50 and standard deviation of 10.
Patient-reported depression as measured by the Patient Reported Outcome Measurement Information System (PROMIS) Short Form v1.0 - Depression 4a | 12 months after enrollment
  Patient-reported depression is measured by the PROMIS Short Form v1.0 - Depression 4a. Scores range from 0 to 100, with higher scores indicating greater symptoms. Scores are normalized to a mean of 50 and standard deviation of 10.
Caregiver-reported anxiety as measured by the Patient Reported Outcome Measurement Information System (PROMIS) Short Form v1.0 - Anxiety 4a | 12 months after enrollment
  Caregiver-reported anxiety is measured by the PROMIS Short Form v1.0 - Anxiety 4a. Scores range from 0 to 100, with higher scores indicating greater symptoms. Scores are normalized to a mean of 50 and standard deviation of 10.
Caregiver-reported depression as measured by the Patient Reported Outcome Measurement Information System (PROMIS) Short Form v1.0 - Depression 4a | 12 months after enrollment
  Caregiver-reported depression is measured by the PROMIS Short Form v1.0 - Depression 4a. Scores range from 0 to 100, with higher scores indicating greater symptoms. Scores are normalized to a mean of 50 and standard deviation of 10.
Patient-reported generic quality of life as measured by the EuroQoL EQ-5D-5L | 12 months after enrollment
  Patient-reported generic quality of life is measured by the EQ-5D. Scores range from 0 to 1, with higher scores indicating better health.
Caregiver-reported generic quality of life as measured by the EuroQoL EQ-5D-5L | 12 months after enrollment
  Caregiver-reported generic quality of life is measured by the EQ-5D. Scores range from 0 to 1, with higher scores indicating better health.
Patient progression-free survival | 12 months after diagnosis of recurrent high-grade non-muscle invasive bladder cancer, up to 12 months post enrollment
  The evaluation of the effect of treatment choice on progression-free survival. Survival times are calculated from the date of diagnosis of recurrent high-grade non-muscle invasive bladder cancer to the event (metastasis or death). A progression is defined as any subsequent episode of muscle-invasive (T2-T4) disease in the bladder or elsewhere in the urinary tract AND/OR locoregional (true pelvic/common iliac) nodal disease (N+) AND/OR distant metastasis (M+) (for cystectomy arm this includes findings at cystectomy). Censoring occurs at the last electronic health record review or death.
Patient bladder cancer-specific survival | 12 months after diagnosis of recurrent high-grade non-muscle invasive bladder cancer, up to 12 months post enrollment
  The evaluation of the effect of treatment choice on bladder cancer-specific survival. Survival times are calculated from the date of diagnosis of recurrent high-grade non-muscle invasive bladder cancer to the event (death from bladder cancer). Censoring occurs at the last electronic health record review or date of death from bladder cancer.

CONTACTS AND LOCATIONS:
Overall Officials: John L Gore, MD, MS, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (6):
- United States (6):
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - University of Iowa, Iowa City, Iowa
  - University of North Carolina, Chapel Hill, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No